CLINICAL TRIAL: NCT01800877
Title: Optimal Vasopressor Titration Pilot Randomized Controlled Trial
Acronym: OVATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francois Lamontagne (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor-Investigator, Francois Lamontagne, Assistant Professor, Universite de Sherbrooke, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVATION
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Hypotension; Shock
Keywords: hypotension; vasopressors; titration; tissue perfusion; organ failure
MeSH Terms: conditions — Hypotension; Shock | interventions — Vasoconstrictor Agents; Phenylephrine; Dopamine; Norepinephrine; Epinephrine; Vasopressins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal Approach (Other): In the liberal approach group, we will titrate vasopressors to maintain mean arterial pressures between 75 and 80 mmHg.
  Interventions: Drug: Vasopressors
- Restrictive Approach (Other): We will titrate vasopressors to maintain mean arterial pressures between 60 and 65 mmHg.
  Interventions: Drug: Vasopressors

INTERVENTIONS:
Drug: Vasopressors
  Other Names: phenylephrine; dopamine; norepinephrine; epinephrine; vasopressin

SUMMARY:
The purpose of this research study is to determine if it is better to give vasopressors to patients to maintain a higher blood pressure target versus a lower blood pressure target. This study is important because the information we find out will help us know how best to administer vasopressors in patients with shock in the ICU.

DETAILED DESCRIPTION:
Patients who are admitted to the intensive care unit (ICU) commonly suffer from shock, a condition that causes life-threatening low blood pressure. Low blood pressure makes it difficult for the body to deliver blood to all of its organs. The standard treatment doctors in the ICU use for their patients is to give medications that help increase blood pressure. These medications are called vasopressors. There can be side effects related to using vasopressors. The purpose of this research study is to determine if it is better to give vasopressors to patients to maintain a higher blood pressure target versus a lower blood pressure target. This study is important because the information we find out will help us know how best to administer vasopressors in patients with shock in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Who are receiving vasopressors for distributive shock
2. Who are older than 16 years of age at the time of eligibility.
3. Who are under the direct care of the ICU team regardless of location.
4. Who have received a minimum of 30 mL/kg of intravenous fluids (2100 mL for a 70 kg patient) before enrolment OR the most responsible physician has good reasons to believe that more fluid resuscitation is no longer required and could be harmful.
5. Who the treating physician believes will need vasopressors for at least 6 hours once enrolled.

Exclusion Criteria:

1. Have received vasopressors for more than 24 consecutive hours; if vasopressors are discontinued for >= 2 hours then restarting vasopressors will constitute a distinct vasopressor episode and the clock will be reset.
2. Are judged by the treating physician to be in obvious cardiogenic shock after an acute myocardial infarction (based on new ST segment elevations on ECG or obvious echocardiographic findings).
3. Have obvious haemorrhagic shock as a consequence of a clearly identified source of blood loss.
4. Require vasopressors after cardiac surgery as a result of cardiopulmonary bypass-induced hypotension.
5. Who have a specific indication for catecholamine therapy other than shock (i.e. angioedema or intracranial hypertension).
6. If the attending team has agreed to withhold or withdraw life sustaining care.
7. Concurrent enrollment in interventional trials that do not meet guidelines (see ccctg.ca) for co-enrollment (co-enrollment is permissible if there is no potential interaction between the protocols; this will be addressed case by case).
8. Prior randomization in this study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lamontagne, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (10):
- Mercy Hospital, St Louis, Missouri, United States
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - Queens Elizabeth II Hospital, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Mt Sinai Hospital, Toronto, Ontario
  - Sunnybrooke HSC, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Hopital L'Enfant-Jesus, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2013 to August 2014, intensive care units (ICUs) at 11 academic hospitals in Canada and the USA participated in this open-label randomized controlled trial with approval from their local research ethics boards.
Groups:
- Liberal Approach: In the liberal approach group, we will titrate vasopressors to maintain mean arterial pressures between 75 and 80 mmHg.
  Vasopressors
- Restrictive Approach: We will titrate vasopressors to maintain mean arterial pressures between 60 and 65 mmHg.
  Vasopressors
Period: Overall Study
Arm/Group | Liberal Approach | Restrictive Approach
Started | 60 | 60
Completed | 58 | 60
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal Approach | Restrictive Approach | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (13) | 66 (13) | 65 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 35 | 31 | 66
Region of Enrollment [Number; unit: participants]
  Canada | 57 | 57 | 114
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: MAP While on Vasopressors
Description: The primary feasibility outcome will be the difference in the means of mean arterial pressures (MAP) while on vasopressors and we define acceptable adherence (the threshold for feasibility) by a difference of at least 5 mmHg while on vasopressors (rejecting the null hypothesis of a difference of less than 5 mmHg - see proposed sample size).
Time Frame: While on vasopressors from randomization until 28 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Liberal Approach | Restrictive Approach
Number analyzed (Participants) | 58 | 60
mmHg | 79 (5) | 70 (5)

ADVERSE EVENTS:
Arm/Group | Liberal Approach | Restrictive Approach
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 45/60 | 41/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal Approach (N=60) | Restrictive Approach (N=60)
Cardiac arrythmia (Cardiac disorders) | 21 (22) | 12 (13)
Myocardial injury (Cardiac disorders) | 9 (9) | 11 (11)
Bowel ischemia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Digit or limb necrosis (Vascular disorders) | 1 (1) | 3 (3)
Gastric feeding intolerance (Gastrointestinal disorders) | 7 (7) | 6 (6)
Venous thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)
Major bleeding (Blood and lymphatic system disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes